CLINICAL TRIAL: NCT03703440
Title: Evaluation of a Group Education Program to Improve the Transition From Pediatric to Adult Care for Emerging Adults With Type 1 Diabetes
Brief Title: Group Education Trial to Improve Transition in Type 1 Diabetes
Acronym: GET-IT-T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: St. Justine's Hospital (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Meranda Nakhla, Assistant Professor, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MP-37-2019-4434
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 1; Type1diabetes; Insulin Dependent Diabetes
Keywords: Transition care; Pediatric; Adolescent; Education; Hemaglobin A1c; Health Services; Randomized Controlled Trial
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Active arm: Patients randomized to the active arm will be asked to attend ≥ 3 group education sessions, in addition to their usual diabetes clinic visits every 3 months, over the 12-month intervention period. Group education sessions will coincide with regularly scheduled clinic visits.
  Control arm: Patients randomized to usual care will attend their usual 3-month interval diabetes clinic visits, over the 12-month intervention period, which consists of visits with their diabetes care physician.
Who Masked: Outcomes Assessor
Masking Description: Data analysts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): ≥3 group education sessions (60 minutes per session) in addition to usual diabetes care, every 3 months for 12 months. Each group session (3-8 patients per group) will be facilitated by a diabetes nurse educator and/or dietitian. The group session content will be guided by the needs of the group participants. The group discussion will end with participants setting goals for their next appointment.
  Interventions: Other: Active arm
- Control (Other): Usual diabetes care, every 3 months for 12 months, which consists of visits with their diabetes care physician. In addition, as per usual diabetes care, an individual education session and written information will be provided before formal transfer.
  Interventions: Other: Control arm

INTERVENTIONS:
Other: Active arm — ≥3 group education sessions in addition to usual diabetes care, every 3 months for 12 months
  Arms: Active
Other: Control arm — Usual diabetes care, every 3-month for 12 months
  Arms: Control

SUMMARY:
The investigators will conduct a randomized controlled trial (RCT) to examine group education visits as an innovative and potentially cost-effective approach to transition care delivery, that can be easily integrated into usual diabetes care. Among emerging adults with type 1 diabetes (T1D), the investigators aim to assess the effect of group education visits integrated into pediatric care, compared with usual care on Hemoglobin A1c (HbA1c), adverse outcomes and psychosocial measures after the transfer to adult care. The investigators will conduct a multi-site, parallel group, blinded (outcome assessors, data analysts), superiority Randomized Controlled Trial (RCT) of adolescents with T1D (17 years of age) followed at one of the two university teaching hospital-based pediatric diabetes clinics in Montreal. Interventions will occur over 12-months. Follow-up will be to 24 months from enrollment.

DETAILED DESCRIPTION:
Rationale. The transition from pediatric to adult diabetes care is a challenging period for adolescents and emerging adults (ages 18-30 years) with type 1 diabetes (T1D). It is characterized by a deterioration in glycemic control (Hemoglobin A1c [HbA1c]), decreased adherence to self-management tasks and to clinic attendance and an increased risk of adverse outcomes. The investigators propose to examine group education visits as a potentially cost-effective approach. In emerging adults with T1D, the investigators hypothesize that group education visits, as compared with usual care, will result in better HbA1c, less adverse outcomes and better psychosocial outcomes after the transfer to adult care.

Primary Aim. To determine the impact of group educations visits, compared with usual care, on HbA1c after the transfer to adult care.

Secondary Aims. 1. To determine the impact of group education visits, compared with usual care, on time between last pediatric and first adult T1D visit (gap > 6 months), emergency department (ED) visits and hospitalizations, severe hypoglycemic events, stigma, self-efficacy, disease knowledge, transition readiness, quality of life (QOL) and diabetes distress, after the transfer to adult care. 2. To determine the cost-effectiveness of group education visits.

Methods. The investigators will conduct a multi-site, parallel group, blinded (outcome assessors, data analysts), superiority Randomized Controlled Trial (RCT) of adolescents with T1D (17 years of age) followed at one of the two university teaching hospital-based pediatric diabetes clinics in Montreal. Patients will be recruited over 24 months. Interventions will occur over 12-months. Follow-up will be to 24 months from enrollment. Allocation will be concealed with a 1:1 intervention to control ratio . Visits in the active arm will consist of a group education session followed by an individual appointment with the diabetes care physician every 3-months. The group education session, facilitated by a diabetes nurse educator or dietitian, will consist of a patient-driven discussion on topics relevant to adolescents with T1D. Patients in the control group, will have in parallel with the intervention group, individual appointments with their diabetes provider as per usual care. The primary outcome is the change in HbA1c measured at 24 months (HbA1c measured at 24 months - HbA1c measured at baseline). Secondary outcomes are delays in establishing adult T1D care (Y/N), T1D-related hospitalizations and ED-visits (rates/P-Y), severe hypoglycemic events, stigma, self-efficacy, diabetes knowledge, transition readiness, diabetes distress, and QOL. Assessments are at baseline, 12 and 24 months . Analysis will be by intention to treat. Outcomes will be calculated and compared between the two trial arms using differences with 95% Confidence Intervals, along with a cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with a diagnosis of Type 1 Diabetes
* 16 to 17 years of age
* Receiving diabetes care at one of two university teaching hospital-based pediatric diabetes clinics in Montreal: Montreal Children's Hospital (MCH) or Centre Hospitalier Universitaire Sainte Justine (CHUSJ)
* Fluent in English or French

Exclusion Criteria:

* Severe neurocognitive disabilities that may preclude patient's ability to participate in a group education visit
* Patients with conditions associated with shortened erythrocyte survival, such as hemolytic anemia or other conditions associated with inaccurate HbA1c

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Hemaglobin A1c (HbA1c) | 0, 12, 24 months
  HbA1c will be measured using an A1c Test Kit, which is a non-fasting, finger stick, whole blood test

SECONDARY OUTCOMES:
Delay in establishing adult Diabetes Care (gap in care>6 months) | 24 months
  Delay greater than 6 months (Y/N) between the last Diabetes Care visit with a pediatric care physician and the first Diabetes Care visit with an adult care physician will be derived from the Physician Service Claims Database (RAMQ) and medical record chart
Delay in establishing adult Diabetes Care (days) | 24 months
  Time in days between the last Diabetes Care visit with a pediatric care physician and the first Diabetes Care visit with an adult care physician will be derived from the Physician Service Claims Database (RAMQ) and medical record chart
Diabetes-related hospitalizations | 0, 12, 24 months
  Any diabetes-related hospitalizations in the past 12 months, expressed as number of hospitalizations per person-years (P-Y) at risk will be derived from the Hospital Discharge Database (Med-Echo) and medical record chart
Diabetes-related emergency department visits | 0, 12, 24 months
  Any diabetes-related emergency-department visits in the past 12 months, expressed as number of emergency department visits per person-years (P-Y) at risk will be derived from the Physician Service Claims Database (RAMQ) and medical record chart
Severe hypoglycemic events | 0,12, 24 months
  Any patient-reported severe hypoglycemic events in the past 12 months
Stigma | 0,12, 24 months
  Presence of stigma defined as an affirmative response to at least one of 3 key items on the Barriers to Diabetes Adherence in Adolescence (BDA) questionnaire stigma subscale (score >2 on a 5-point Likert-type scale)
Self-efficacy | 0,12, 24 months
  Self-efficacy for Diabetes Self-Management Measure (SEDM) assesses self-efficacy. The score ranges from 1 to 10. All item scores are averaged to compute the score. A higher score represents a better outcome.
Diabetes knowledge | 0, 12, 24 months
  L'Aide aux Jeunes Diabétiques Diabetes Knowledge and Skills Questionnaire assesses diabetes knowledge. The score ranges from 0 to 50. The number of correct items are summed to compute the score. A higher score represents a better outcome.
Transition readiness | 0, 12 months
  Am I ON TRAC? For Adult Care Questionnaire (Youth Version of Questionnaire) measures transition readiness. Scores range from 13 to 64 on the Knowledge Scale. Item scores are summed to compute the Knowledge Scale score. Higher scores on the Knowledge Scale represent a better outcome. Raw scores range from 8 to 45 on the Behaviour Index. Item scores are summed to compute the raw scores on the Behaviour Index. Higher raw scores on the Behaviour Index represent a better outcome. Cut-off scores range from 0 to 9 on the Behaviour Index. Threshold scores are summed to compute the cut-off scores on the Behaviour Index. Higher cut-off scores on the Behaviour Index represent a better outcome.
Diabetes distress | 0, 12, 24 months
  Diabetes Distress Scale for Adults with Type 1 Diabetes (T1-DDS) measures diabetes-related distress. The Total Score ranges from 1 to 6. All item scores are averaged to compute the Total Score. A higher Total Score represents a worse outcome. Scores range from 1 to 6 on the 7 Subscales (1. Powerlessness, 2. Management Distress, 3. Hypoglycemia Distress, 4. Negative Social Perceptions, 5. Eating Distress, 6. Physician Distress, 7. Friend/Family Distress) and Screener. Item scores are averaged to compute the Subscale and Screener scores. Higher Subscale and Screener scores represent a worse outcome.
Quality of life (Generic Core) | 0, 12, 24 months
  Pediatric Quality of Life Inventory (PedsQL) Generic Core Scale assesses Health-Related Quality of Life. Scores are transformed on a scale from 0 to 100. The Scale Scores (Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning) range from 0 to 100. To create Scale Scores, the mean is computed as the sum of the items over the number of items answered. Higher Scale Scores represent a better outcome. To create the Psychosocial Health Summary Score, the mean is computed as the sum of the items over the number of items answered in the Emotional, Social, and School Functioning Scales. The Physical Health Summary Score is the same as the Physical Functioning Scale Score. The Total Scale Score ranges from 0 to 100. To create the Total Scale Score, the mean is computed as the sum of all the items over the number of items answered on all the Scales. A higher Total Scale Score represents a better outcome.
Quality of life (Diabetes Module) | 0, 12, 24 months
  Pediatric Quality of Life Inventory (PedsQL) Diabetes Module assesses diabetes-specific quality of life. Scores are transformed on a scale from 0 to 100. The Scale Scores by Dimension (About My Diabetes, Treatment-I, Treatment II, Worry, and Communication) range from 0 to 100. To calculate Scale Scores by Dimension, the mean is computed as the sum of the items over the number of items answered. Higher Scale Scores represent a better outcome. To calculate the Total Score, the mean is computed as the sum of all the items over the number of items answered on all the Scales. A higher Total Score represents a better outcome.
Cost effectiveness (HbA1c) | 12 and 24 months
  Cost-effectiveness of group education visits compared with usual care in terms of incremental cost effectiveness ratio (ICER) for HbA1c
Cost effectiveness (QOL) | 12 and 24 months
  Cost-effectiveness of group education visits compared with usual care in terms of incremental cost effectiveness ratio (ICER) for QOL
Cost effectiveness (self-efficacy) | 12 and 24 months
  Cost-effectiveness of group education visits compared with usual care in terms of incremental cost effectiveness ratio (ICER) for self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Meranda Nakhla, MD, MSc, Principal Investigator — Montreal Children's Hospital - McGill University Health Centre (MUHC)
Locations (2):
- Canada (2):
  - Centre Hospitalier Universitaire Sainte-Justine (CHUSJ), Montreal, Quebec
  - Montreal Children's Hospital - McGill University Health Centre (MUHC), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data supporting the results reported in the published research articles, after de-identification will be available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available immediately following article publication and ending 5 years after article publication.
Access Criteria: Data will be shared with researchers who provide a scientifically sound proposal that has been approved by an independent Institutional Review Board and for analyses that addresses the aims specified in the proposal (e.g. for individual participant data meta-analysis). Proposals should be submitted to meranda.nakhla@mcgill.ca. Data requestors will need to sign a data access agreement. Data will be available up to 5 years following article publication at (Link to be included).

REFERENCES:
- [Background] Brazeau AS, Nakhla M, Wright M, Henderson M, Panagiotopoulos C, Pacaud D, Kearns P, Rahme E, Da Costa D, Dasgupta K. Stigma and Its Association With Glycemic Control and Hypoglycemia in Adolescents and Young Adults With Type 1 Diabetes: Cross-Sectional Study. J Med Internet Res. 2018 Apr 20;20(4):e151. doi: 10.2196/jmir.9432. PMID 29678801
- [Background] Diabetes Canada Clinical Practice Guidelines Expert Committee; Wherrett DK, Ho J, Huot C, Legault L, Nakhla M, Rosolowsky E. Type 1 Diabetes in Children and Adolescents. Can J Diabetes. 2018 Apr;42 Suppl 1:S234-S246. doi: 10.1016/j.jcjd.2017.10.036. No abstract available. PMID 29650103
- [Background] Nakhla M, Rahme E, Simard M, Larocque I, Legault L, Li P. Risk of ketoacidosis in children at the time of diabetes mellitus diagnosis by primary caregiver status: a population-based retrospective cohort study. CMAJ. 2018 Apr 9;190(14):E416-E421. doi: 10.1503/cmaj.170676. PMID 29632036
- [Background] Michaud S, Dasgupta K, Bell L, Yale JF, Anjachak N, Wafa S, Nakhla M. Adult care providers' perspectives on the transition to adult care for emerging adults with Type 1 diabetes: a cross-sectional survey. Diabet Med. 2018 Jul;35(7):846-854. doi: 10.1111/dme.13627. Epub 2018 May 2. PMID 29577410
- [Background] Nakhla M, Bell LE, Wafa S, Dasgupta K. Improving the transition from pediatric to adult diabetes care: the pediatric care provider's perspective in Quebec, Canada. BMJ Open Diabetes Res Care. 2017 Jun 30;5(1):e000390. doi: 10.1136/bmjdrc-2017-000390. eCollection 2017. PMID 28761657
- [Background] Nakhla M, Rahme E, Simard M, Guttmann A. Outcomes associated with a pediatric clinical diabetes network in Ontario: a population-based time-trend analysis. CMAJ Open. 2017 Jul 24;5(3):E586-E593. doi: 10.9778/cmajo.20170022. PMID 28747349
- [Background] Brazeau AS, Nakhla M, Wright M, Panagiotopoulos C, Pacaud D, Henderson M, Rahme E, Da Costa D, Dasgupta K. Stigma and Its Impact on Glucose Control Among Youth With Diabetes: Protocol for a Canada-Wide Study. JMIR Res Protoc. 2016 Dec 15;5(4):e242. doi: 10.2196/resprot.6629. PMID 27979791
- [Background] Wafa S, Nakhla M. Improving the Transition from Pediatric to Adult Diabetes Healthcare: A Literature Review. Can J Diabetes. 2015 Dec;39(6):520-8. doi: 10.1016/j.jcjd.2015.08.003. Epub 2015 Oct 20. PMID 26498219
- [Background] Jefferies CA, Nakhla M, Derraik JG, Gunn AJ, Daneman D, Cutfield WS. Preventing Diabetic Ketoacidosis. Pediatr Clin North Am. 2015 Aug;62(4):857-71. doi: 10.1016/j.pcl.2015.04.002. Epub 2015 May 30. PMID 26210621
- [Background] Nakhla M, Daneman D, To T, Paradis G, Guttmann A. Transition to adult care for youths with diabetes mellitus: findings from a Universal Health Care System. Pediatrics. 2009 Dec;124(6):e1134-41. doi: 10.1542/peds.2009-0041. Epub 2009 Nov 23. PMID 19933731
- [Background] Guttmann A, Nakhla M, Henderson M, To T, Daneman D, Cauch-Dudek K, Wang X, Lam K, Hux J. Validation of a health administrative data algorithm for assessing the epidemiology of diabetes in Canadian children. Pediatr Diabetes. 2010 Mar;11(2):122-8. doi: 10.1111/j.1399-5448.2009.00539.x. Epub 2009 Jun 5. PMID 19500278
- [Background] Nakhla M, Daneman D, Frank M, Guttmann A. Translating transition: a critical review of the diabetes literature. J Pediatr Endocrinol Metab. 2008 Jun;21(6):507-16. PMID 18717235
- [Derived] Mok E, Henderson M, Dasgupta K, Rahme E, Hajizadeh M, Bell L, Prevost M, Frei J, Nakhla M. Group education for adolescents with type 1 diabetes during transition from paediatric to adult care: study protocol for a multisite, randomised controlled, superiority trial (GET-IT-T1D). BMJ Open. 2019 Nov 11;9(11):e033806. doi: 10.1136/bmjopen-2019-033806. PMID 31719096